CLINICAL TRIAL: NCT04843111
Title: The MenQuadfi® Pregnancy Registry: A Surveillance Registry to Assess the Safety of MenQuadfi® Among Exposed Pregnant Women and Their Offspring
Brief Title: Observational, Passive Surveillance Program to Collect Information on Women and Their Offspring Exposed to MenQuadfi® During Pregnancy, in United States (US)
Status: Recruiting | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: MEQ00070; U1111-1250-2672 (Registry Identifier: ICTRP); MEQ00070 (Other: Sanofi Identifier)
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Meningococcal Infection
MeSH Terms: conditions — Meningococcal Infections | interventions — Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 22 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women and their offspring(s): Pregnant women and their offspring(s) exposed to MenQuadfi® during their pregnancy or within 30 days prior to their LMP
  Interventions: Biological: Meningococcal polysaccharide (serogroups A, C, Y, and W) tetanus toxoid conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal polysaccharide (serogroups A, C, Y, and W) tetanus toxoid conjugate vaccine — Pharmaceutical form: Solution for injection Route of administration: Intramuscular
  Other Names: Meningococcal A-C-Y-W135 (T CONJ) vaccine

SUMMARY:
Primary Objective:

To assess maternal, obstetrical, pregnancy, and neonatal and infant outcomes among women vaccinated with MenQuadfi® during pregnancy or in the 30 days preceding their Last Menstrual Period (LMP).

DETAILED DESCRIPTION:
This study is a prospective pregnancy registry to collect and analyze the outcome of exposure to MenQuadfi™ during pregnancy or within 30 days prior to their LMP. The registry will encourage prospective registration, which is defined as registration of a pregnancy exposure prior to knowledge or perceived knowledge of the pregnancy outcome.

Exposed pregnant women will be followed up to the end of their pregnancy, and the offspring(s) will be followed up to 1 year of age.

ELIGIBILITY:
Inclusion Criteria:

The eligible population will include pregnant women and their offspring residing in the US and its territories who are exposed to MenQuadfi® during their pregnancy or within 30 days prior to their LMP, for whom the exposure is reported to the pregnancy registry.

Reports of MenQuadfi® pregnancy exposure must contain the following information:

* Sufficient evidence to confirm that vaccination occurred during the pregnancy or in the 30 days preceding the LMP;
* Vaccine name (brand or generic) is provided (i.e., MenQuadfi®, Meningococcal vaccine, MenACWY conjugate vaccine), or not specified (eg, meningococcal vaccine from an unknown manufacturer).

Exclusion Criteria:

Only post-marketing spontaneous case reports will be included; reports from clinical trials will not be part of the registry.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women and their offspring residing in the US and its territories who are exposed to MenQuadfi® during their pregnancy or within 30 days prior to their last menstrual period (LMP), for whom the exposure is reported to the pregnancy registry.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2028-05-18 (Estimated); Study Completion 2028-05-18 (Estimated)

PRIMARY OUTCOMES:
Percentage of pregnant women with maternal adverse events (AEs) | From vaccination to end of follow-up (i.e.,up to 22 months after cohort entry)
  Maternal adverse events defined as any reported adverse event (AE), following vaccination of a pregnant woman, occurring independent of the pregnancy (e.g., injection site reactions)
Percentage of pregnant women with obstetrical AEs | From vaccination to 28 days after delivery
  Obstetrical adverse events defined as any reported AE, following vaccination of a pregnant woman, related directly to the pregnancy (e.g., complications of pregnancy, labor and delivery, and puerperium)
Percentage of pregnant women with pregnancy AEs | On day of birth
  Pregnancy adverse events defined as any reported AE, following vaccination of a pregnant woman, related to birth outcomes (e.g., live birth, spontaneous abortion/miscarriage, stillbirth/fetal death)

SECONDARY OUTCOMES:
Percentage of offsprings with adverse neonatal AEs | From day of birth to 28 days post-birth
  Neonatal events defined as any reported AE, following vaccination of a pregnant woman, directly related to the infant and assessed immediately after birth or within the first 28 days of life (e.g., congenital anomalies)
Percentage of offsprings with adverse infant AEs | From day 29 post-birth to 365 days post-birth
  Infant events defined as any reported AE, following vaccination of a pregnant woman, directly related to the infant occurring / diagnosed between days 29 and 365 post-birth

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Pennsylvania Locations, Swiftwater, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org